CLINICAL TRIAL: NCT04077294
Title: Epidemiological Patterns, Management Strategies and Cost Analysis of Care for the Patient With Perioperative Myocardial Injury When BNP is Used as a Screening Tool for Non-Cardiac Surgery
Brief Title: Preoperative BNP: Epidemiological Patterns, Management Strategies and Cost Analysis of Care
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00086046
Record Dates: First submitted 2019-07-05; First posted 2019-09-04 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Myocardial Infarction Postoperative; Myocardial Injury; Death, Cardiac
Keywords: Preoperative BNP; Perioperative cardiac risk stratification; Myocardial injury after non-cardiac surgery (MINS); Canadian Cardiovascular Society (CCS) guidelines
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative BNP used for cardiac risk stratification: Cohort of patients recruited in the pre-admission clinic who qualified for, and underwent, preoperative BNP screening according to CCS guidelines.
  Interventions: Other: Cardiac risk stratification using preoperative BNP measurement, followed by postoperative cardiac monitoring
- Preoperative BNP not used for cardiac risk stratification: Cohort of patients from patient care database (SPOR) who qualified for preoperative BNP screening according to CCS guidelines, but did not receive screening due to surgery occurring before the implementation of the CCS guidelines.
  Interventions: Other: Use of traditional perioperative cardiac risk stratification only

INTERVENTIONS:
Other: Cardiac risk stratification using preoperative BNP measurement, followed by postoperative cardiac monitoring — Patients undergoing non-cardiac surgery risk stratified using BNP measurements according to CCS guidelines.
  Groups: Preoperative BNP used for cardiac risk stratification
Other: Use of traditional perioperative cardiac risk stratification only — Patients undergoing non-cardiac surgery risk stratified using tools other than BNP measurement such as revised cardiac risk index (RCRI).
  Groups: Preoperative BNP not used for cardiac risk stratification

SUMMARY:
Recently, the use of preoperative BNP as a preoperative risk stratifcation tool was added to the Canadian Cardiovascular Society (CCS) guidelines (4) on perioperative cardiac risk assessment and management for patients who undergo noncardiac surgery, based on the prognostic value of preoperative BNP in indentifiy patients at significant risk of 30-day mortality, nonfatal myocardial infarction, or myocardial injury after noncardiac surgery (MINS). While the value of screening for high risk patients through the use of preoperative BNP been demonstrated, the management of postoperative ischemia is less clear. Therefore, this study aims to:

1. Evaluation of the use of BNP as a preoperative screening biomarker; how often is it ordered in Anesthesia Preadmission Clinic and what is the incidence of a positive result (BNP ≥ 92 ng/L)
2. Determine the incidence of myocardial injury after non-cardiac surgery (MINS) at 30 days and myocardial infarction at 1 year at a tertiary care center when BNP is used as a screening tool
3. Record patterns of management of patients with MINS
4. Determine the cost associated with the different patterns of management of MINS
5. Comparison with a cohort group who qualified for BNP screening according to CCS guidelines but did not have it measured. The investigators will attempt to evaluate the cohort group for MINS at 30 days and myocardial infarction at 1 year.

DETAILED DESCRIPTION:
Major cardiac complications are responsible for at least a third of perioperative deaths and are associated with significant morbidity, prolonged hospitalization and increased costs. This number is expected to rise as more surgeries are undertaken in older and frailer patients. The term myocardial injury after noncardiac surgery (MINS) is used to describe all myocardial injury due to ischemia occurring in the first 30 days after surgery. MINS includes:

1. myocardial infarction (cardiac troponin I ≥ 0.04 ug/L) with at least one of: symptoms of ischemia, new ST segment / T wave changes or new left bundle branch block, pathological Q waves, new loss of viable myocardium or regional wall motion abnormality on echocardiogram, intracoronary thrombus identified on angiogram.
2. myocardial injury without MI (elevated troponin without the additional criteria needed to diagnose MI).

The Canadian Cardiovascular Society (CCS) has developed a set of guidelines to help stratify which patients are at higher risk for cardiac mortality. In the latest revision of these guidelines, preoperative B-type natriuretic peptide (BNP) has been identified as a powerful independent predictor of perioperative cardiovascular complications. BNP is a protein released from ventricular cardiomyocytes. It is released in limited amounts during physiological conditions but this is increased significantly in ventricular failure, inflammation, fibrosis, ischemia and hypoxia. Rodseth et al. conducted a systematic review of the prognostic value of preoperative BNP and postoperative BNP in noncardiac surgery and showed that elevated preoperative BNP (i.e. ≥ 92 ng/l) carries a significant risk of 30-day mortality or nonfatal MI (21.8%). This is a significantly lower BNP value compared to what is typically seen in congestive cardiac failure patients. This study has been used to support the most recent CCS guidelines which add preoperative BNP as an important preoperative cardiac risk stratification tool. According to the CCS guidelines, patients with an elevated preoperative BNP should have daily troponins measured for 48 - 72 hours after surgery.

Troponins are components of the myocardial cell involved in contractility, specific subtypes I and T are expressed almost exclusively in the heart. An elevated troponin reflects necrosis of myocardial cells and is extremely useful in the diagnosis of a myocardial infarction. Even a slight elevation in postoperative troponins (TnTi ≥ 0.03ng/ml) without ischemic clinical symptoms can lead to a higher mortality, nonfatal cardiac arrest, nonfatal congestive heart failure, and nonfatal stroke.

While the value of screening for high risk patients through the use of preoperative BNP been demonstrated, the management of postoperative ischemia is less clear. At present, CCS guidelines recommend optimizing aspirin and statin therapy in patients with MINS, but no clear strategy has been elucidated. Evidence to support the use of aspirin and statins comes from the POISE trial. The MANAGE trial recommends starting patients who are not at risk of bleeding on the oral anticoagulant dabigatran for two years. Patients with ST-elevation MI carry a high mortality risk without reperfusion therapy (percutaneous coronary intervention or coronary artery bypass graft) and a high risk of bleeding with it. Patients with non ST-elevation MI may also require revascularization and subsequent dual antiplatelet therapy. It is evident from this brief overview that management of MINS varies from the non-invasive (aspirin and statin administration) to the invasive (PCI or CABG) depending on the extent of myocardial injury, hemodynamic stability and risk of bleeding secondary to the primary surgical procedure.

Screening for patients at risk of MINS by measuring BNP may have a significant impact on health care resources. 80% of patients with MINS are asymptomatic and go unrecognized. Screening for patients who are at risk of postoperative myocardial ischemia will ostensibly uncover a new population of patients i.e. those who, prior to BNP screening, experienced subclinical postoperative ischemia which went undiagnosed until a later juncture by which time potentially worse and irreversible myocardial injury had occurred.

In this study the objectives are to investigate:

1. incidence of qualification for BNP measurement as determined by CCS guidelines
2. incidence of patients with BNP ≥ 92 ng/L
3. incidence of MINS (myocardial infarction and myocardial injury without MI) at 30 days and incidence of myocardial infarction at 1 year after surgery
4. evaluate the management of patients with positive troponin after surgery
5. identify a matched cohort group from the SPOR database
6. compare the incidence and timing of MINS in the BNP group versus that in a matched cohort group who qualified for BNP screening but did not have it done
7. determination of cost of screening, diagnosis and management of MINS and MI for up to 1 year after surgery when BNP is used as a screening tool

In this study, elective patients deemed at risk of a postoperative cardiac event will be monitored, as determined by preoperative BNP measurement, up to 1 year postoperatively. BNP positive patients will be monitored for myocardial injury postoperatively by measuring troponin daily for 72 hours. The incidence of MINS (MI and myocardial injury without MI) in BNP positive patients will be determined. Patients with troponin I ≥ 0.04 ug/L will be referred to the cardiology consult service for further evaluation and management. Subsequent management will be categorized as 1) monitor 2) medical management and 3) revascularization. A cost analysis of the management of all three groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients:

  * ≥ 65 years of age
  * ≥ 18 years of age with a revised cardiac risk index (RCRI) ≥ 1
  * between 45 and 64 years of age with significant cardiovascular disease
* Elective non-cardiac surgery with an overnight hospital stay (minimum 1 day)

Exclusion Criteria:

* Subjects < 18 years of age
* Patient refusal to participate
* Patients undergoing cardiac surgery
* Patients undergoing day surgery (< 1day hospital admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients undergoing elective non-cardiac surgery with an overnight hospital stay meeting one of the following criteria:
  1. age ≥ 65
  2. a revised cardiac risk index (RCRI) ≥ 1 (see Appendix 1)
  3. age 45 - 64 with significant cardiovascular disease*
  Patients will be identified and recruited in the anesthesia preadmission clinic prior to surgery.
  *Known history of coronary artery disease, cerebral vascular disease, peripheral artery disease, congestive heart failure, severe PHTN or a severe obstructive intracardiac abnormality (eg, severe aortic stenosis, severe mitral stenosis, or severe hypertrophic obstructive cardiomyopathy).
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Preoperative Brain natriuretic peptide (BNP) ≥ 92 ng/L | From date of preoperative consultation up to the day of surgery, assessed up to 6 months.
  Number of participants with preoperative BNP ≥ 92 ng/L
Postoperative troponin I ≥ 0.04 ug / L | From the end of the surgical procedure to 72 hours postoperatively
  Incidence of myocardial injury in the early postoperative period after non-cardiac surgery (MINS)
Myocardial injury at 30 days after surgery | 30 days after surgery
  Incidence of myocardial injury 30 days after surgery at risk in patients as determined by preoperative BNP measurement
Myocardial injury 1 year after surgery | 1 year after surgery
  Incidence of myocardial injury 1 year after surgery at risk in patients as determined by preoperative BNP measurement

SECONDARY OUTCOMES:
Observation of management patterns 30 days after surgery in patients with myocardial injury after non-cardiac surgery (MINS) | 30 days after surgery
  The management strategies used to treat patients with MINS will be categorized as 1) monitoring only, 2) medical management, or 3) revascularization. There is no measurement tool or scale. This is an observational component where management of myocardial injury after surgery will be broadly categorized as 1) monitoring only, 2) medical management, or 3) revascularization.
Observation of management patterns 1 year after surgery in patients with myocardial injury after non-cardiac surgery (MINS) | 1 year after surgery
  The management strategies used to treat patients with MINS will be categorized as 1) monitoring only, 2) medical management, or 3) revascularization. There is no measurement tool or scale. This is an observational component where management of myocardial injury after surgery will be broadly categorized as 1) monitoring only, 2) medical management, or 3) revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Dillane, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital Pre-Admission Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Background] Udeh BL, Dalton JE, Hata JS, Udeh CI, Sessler DI. Economic trends from 2003 to 2010 for perioperative myocardial infarction: a retrospective, cohort study. Anesthesiology. 2014 Jul;121(1):36-45. doi: 10.1097/ALN.0000000000000233. PMID 24662375
- [Background] van Waes JA, Nathoe HM, de Graaff JC, Kemperman H, de Borst GJ, Peelen LM, van Klei WA; Cardiac Health After Surgery (CHASE) Investigators. Myocardial injury after noncardiac surgery and its association with short-term mortality. Circulation. 2013 Jun 11;127(23):2264-71. doi: 10.1161/CIRCULATIONAHA.113.002128. Epub 2013 May 10. PMID 23667270
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641
- [Background] Rodseth RN, Biccard BM, Le Manach Y, Sessler DI, Lurati Buse GA, Thabane L, Schutt RC, Bolliger D, Cagini L, Cardinale D, Chong CP, Chu R, Cnotliwy M, Di Somma S, Fahrner R, Lim WK, Mahla E, Manikandan R, Puma F, Pyun WB, Radovic M, Rajagopalan S, Suttie S, Vanniyasingam T, van Gaal WJ, Waliszek M, Devereaux PJ. The prognostic value of pre-operative and post-operative B-type natriuretic peptides in patients undergoing noncardiac surgery: B-type natriuretic peptide and N-terminal fragment of pro-B-type natriuretic peptide: a systematic review and individual patient data meta-analysis. J Am Coll Cardiol. 2014 Jan 21;63(2):170-80. doi: 10.1016/j.jacc.2013.08.1630. Epub 2013 Sep 26. PMID 24076282
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on behalf of the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction. Third universal definition of myocardial infarction. Glob Heart. 2012 Dec;7(4):275-95. doi: 10.1016/j.gheart.2012.08.001. Epub 2012 Sep 26. No abstract available. PMID 25689940
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Background] Devereaux PJ, Duceppe E, Guyatt G, Tandon V, Rodseth R, Biccard BM, Xavier D, Szczeklik W, Meyhoff CS, Vincent J, Franzosi MG, Srinathan SK, Erb J, Magloire P, Neary J, Rao M, Rahate PV, Chaudhry NK, Mayosi B, de Nadal M, Iglesias PP, Berwanger O, Villar JC, Botto F, Eikelboom JW, Sessler DI, Kearon C, Pettit S, Sharma M, Connolly SJ, Bangdiwala SI, Rao-Melacini P, Hoeft A, Yusuf S; MANAGE Investigators. Dabigatran in patients with myocardial injury after non-cardiac surgery (MANAGE): an international, randomised, placebo-controlled trial. Lancet. 2018 Jun 9;391(10137):2325-2334. doi: 10.1016/S0140-6736(18)30832-8. PMID 29900874
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280